CLINICAL TRIAL: NCT02598440
Title: A Randomized, Open-Label, Muti-Center Study to Investigate Patient Preference on Dosing in Women With Postmenopausal Osteoporosis Treated With Once-Monthly Ibandronate and Once-Weekly Alendronate. A Six Month, Two-Sequence, and Two-Period Crossover Study
Brief Title: A Study of Ibandronate (Bonviva) in Patients With Post-Menopausal Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MA17843
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Alendronate; Ibandronic Acid

ARMS (2):
- Group A: Ibandronate Then Alendronate (Experimental): Participants wil receive once-monthly oral ibandronate (150 mg tablet) for 3 months followed by and once-weekly oral alendronate (70 mg tablet) in crossover design for 12 weeks.
  Interventions: Drug: Alendronate; Drug: Ibandronate
- Group B: Alendronate Then Ibandronate (Experimental): Participants will receive once-weekly oral alendronate (70 mg tablet) for 12 weeks followed by once-monthly oral ibandronate (150 mg tablet) for 3 months.
  Interventions: Drug: Alendronate; Drug: Ibandronate

INTERVENTIONS:
Drug: Alendronate — Participants wil receive once-weekly oral alendronate (70 mg tablet)
Drug: Ibandronate — Participants wil receive once-monthly oral ibandronate (150 mg tablet)
  Other Names: Bonviva

SUMMARY:
This study will evaluate participant-reported preference for either ibandronate or a comparator drug in women with postmenopausal osteoporosis. The anticipated time of study treatment is 6 months, and the target sample size is 338 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory women
* Diagnosis of post-menopausal osteoporosis
* Women who have never received bisphosphonate therapy, or who have discontinued daily bisphosphonates at least 3 months prior to study entry

Exclusion Criteria:

* Inability to stand or sit in the upright position for greater than or equal to 60 minutes
* Allergy to bisphosphonates;
* Previous or current treatment with weekly or monthly bisphosphonates, or daily bisphosphonates for the last 3 months prior to study entry

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2004-03; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Percentage of participants preferring once-monthly dosing of ibandronate over once-weekly dosing of alendronate | Up to 6 months

SECONDARY OUTCOMES:
Percentage of participants perceiving the once-monthly dosing of ibandronate to be more convenient over once-weekly dosing of alendronate. | Up to 6 months
Incidence of adverse events | Up to approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (50):
- United States (50):
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Tempe, Arizona
  - Laguna Woods, California
  - Mission Viejo, California
  - Oceanside, California
  - San Diego, California
  - Santa Clarita, California
  - Upland, California
  - Vista, California
  - Denver, Colorado
  - Cromwell, Connecticut
  - Waterbury, Connecticut
  - Newark, Delaware
  - Aventura, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Augusta, Georgia
  - Decatur, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - South Bend, Indiana
  - Des Moines, Iowa
  - Wichita, Kansas
  - Bangor, Maine
  - Baltimore, Maryland
  - Worcester, Massachusetts
  - Florissant, Missouri
  - St Louis, Missouri
  - Reno, Nevada
  - Princeton, New Jersey
  - Toms River, New Jersey
  - Orchard Park, New York
  - Raleigh, North Carolina
  - Eugene, Oregon
  - Duncansville, Pennsylvania
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wyomissing, Pennsylvania
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Newport News, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Madison, Wisconsin